CLINICAL TRIAL: NCT05480384
Title: BrUOG 413: A Phase II Study of Adjuvant Trastuzumab Deruxtecan (Enhertu) + Nivolumab For Patients Who Are Disease Free After Completion of Trimodality Treatment For HER-2-Positive Cancers of the Esophagus and Gastroesophageal Junction
Brief Title: Adjuvant Trastuzumab Deruxtecan (Enhertu) & Nivolumab For Patients Who Are Disease Free After Completion of Trimodality Treatment For HER-2+ Cancers of Esophagus & Gastroesophageal Junction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 413
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Adenocarcinoma; Esophageal Cancer; HER-2 Protein Overexpression; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Nivolumab; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Starting Trastuzumab Deruxtecan Dose (Experimental): Trastuzumab deruxtecan, 6.4 mg/kg IV every 3 weeks for 17 doses (12 months)
  Interventions: Drug: Nivolumab; Drug: Trastuzumab deruxtecan
- First Trastuzumab Deruxtecan Dose Reduction (Experimental): Trastuzumab deruxtecan, 5.4 mg/kg IV every 3 weeks for 17 doses (12 months)
  Interventions: Drug: Nivolumab; Drug: Trastuzumab deruxtecan
- Second Trastuzumab Deruxtecan Dose Reduction (Experimental): Trastuzumab deruxtecan, 4.4 mg/kg IV every 3 weeks for 17 doses (12 months)
  Interventions: Drug: Nivolumab; Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Nivolumab — Nivolumab, 360 mg IV every 3 weeks for 17 doses (12 months)
  Other Names: OPDIVO
Drug: Trastuzumab deruxtecan — Given in combination with Nivolumab.
  Other Names: ENHERTU

SUMMARY:
An open label phase II study to determine the safety and preliminary efficacy of the combination of 1-year of adjuvant trastuzumab deruxtecan and nivolumab for patients with HER2 overexpressing esophagogastric adenocarcinoma who have completed chemoradiation followed by esophagectomy.

DETAILED DESCRIPTION:
This is an open label phase II study to determine the safety and preliminary efficacy of the combination of 1-year of adjuvant trastuzumab deruxtecan and nivolumab for patients with HER2 overexpressing esophagogastric adenocarcinoma who have completed chemoradiation followed by esophagectomy. All patients will receive trastuzumab deruxtecan, 6.4 mg/kg IV, and nivolumab, 360 mg IV, every 21 days, for 17 doses over 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed primary adenocarcinoma of the esophagus, esophagogastric junction or (Stomach involvement is allowed.).
2. HER2 overexpression defined by immunohistochemistry (IHC) 3+ or HER2 amplification by fluorescence in situ hybridization (FISH). This may be defined by local or commercial laboratories
3. Completed trimodality treatment with chemoradiation followed by esophagectomy and had an R0 resection but did not achieve a complete pathologic response.
4. 4 - 12 weeks after esophagectomy.
5. Prior to trimodality treatment had stage T1N1-2 M0, T2-3N0-2 M0 disease.
6. Age ≥ 18
7. ECOG performance status 0-1
8. For women of childbearing potential, a negative serum pregnancy test within 7 days prior to registration
9. Women of childbearing potential and male participants must practice highly effective form of non-hormonal contraception throughout the study, which is defined as from study screening (ICF) through 2 months post last treatment; Non-sterilised male partners of a woman of childbearing potential must use a male condom plus spermicide (condom alone in countries where spermicides are not approved) throughout this period.
10. Ability to understand and the willingness to sign a written informed consent document.
11. LVEF ≥ 50% within 28 days before randomization/enrollment.
12. Adequate organ and bone marrow function within 14 days before randomization/enrolment. All parameters must meet the inclusion criteria on the same day, and must be the most recent results available.
13. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of treatment. Women of childbearing potential are defined as those who are not surgically sterile (i.e. underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
14. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, from the time of screening and must agree to continue using such precautions for 7 months after the last dose of treatment. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of treatment. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
15. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of treatment. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of enrollment, throughout the study and for 4 months after the last dose of treatment. Preservation of sperm should be considered prior to enrollment in this study.
16. Female subjects must not donate, or retrieve for their own use, ova from the time of enrollment and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrollment in this study.

Exclusion Criteria:

1. Has substance abuse or any other medical conditions such as clinically significant cardiac or psychological conditions, that may, in the opinion of the investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
2. Patients with a medical history of myocardial infarction (MI) within 6 months before enrollment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.
3. Corrected QT interval (QTcF) prolongation to > 470 msec (females) or >450 msec (males) based on average of the screening triplicate12-lead ECG.
4. History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.
5. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.

   * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
   * Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the eCRF for patients who are included in the study.
   * Prior pneumonectomy (complete)
6. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
7. Active primary immunodeficiency, known uncontrolled active HIV infection or active hepatitis B or C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1. Subjects with past or resolved hepatitis B virus (HBV) infection who are anti-HBc positive (+) are eligible only if they are HBsAg negative (-).
8. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
9. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of trastuzumab deruxtecan. Note: Patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of treatment.
10. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline. Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to [randomization/enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:

    * Chemotherapy-induced neuropathy
    * Fatigue
11. Known allergy or hypersensitivity to study treatment or any of the study drug excipients.
12. History of severe hypersensitivity reactions to other monoclonal antibodies.
13. Pregnant or breastfeeding female patients, or patients who are planning to become pregnant.
14. Multiple primary malignancies within 3 years, with the exception of

    * adequately resected non-melanoma skin cancer
    * curatively treated in-situ disease
    * other solid tumors curatively treated
    * contralateral breast cancer.
15. A pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or pleurx catheter
16. No prior treatment with nivolumab, other immunotherapy agents for esophageal cancer, or trastuzumab deruxtecan or other HER2 directed agent or other investigational anti-cancer agent.
17. Pregnant women, or patients planning to become pregnant, are excluded from this study because both nivolumab and trastuzumab deruxtecan have the potential for teratogenic or abortifacient effects.
18. In order for patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) to be eligible, they must be on a stable highly active antiretroviral therapy (HAART) regimen, have CD4 counts > 350, with no detectable viral load on quantitative PCR within 4 weeks of registration.
19. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease, Crohn's, ulcerative colitis, and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patient with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment (which would preclude them) but should otherwise be eligible. All information to be documented by treating physician.
20. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement (such as Hashimoto's thyroiditis), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event), as confirmed by treating physician.
21. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of day 1 study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
22. Any other medical condition that will prevent the safe administration of study drugs in the opinion of the treating physician.
23. Planned concomitant, non-protocol directed anti-cancer therapy during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety of the addition of adjuvant trastuzumab deruxtecan with nivolumab for patients with esophagogastric cancer who have completed trimodality treatment | First dose of study treatment, through 30-days post last dose of drug, approximately 13 months
  Measured by the rates of clinically significant treatment-related grade ≥3 adverse events or pneumonitis.

SECONDARY OUTCOMES:
Disease-free survival with adjuvant trastuzumab deruxtecan & nivolumab after completion of trimodality treatment for HER2+ esophageal cancer. | First dose of study treatment until time of cancer recurrence or death from any cause, whichever occurs first, maximum of 36 months
  Participants alive without disease recurrence are censored at date of last disease evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Principal Investigator — Lifespan Cancer Institute; Manish A Shah, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Weill Cornell Medicine/New York-Presbyterian, New York, New York
  - Lifespan Cancer Institute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No